CLINICAL TRIAL: NCT01585883
Title: A Pilot Trial of a Self-Management Intervention for Breathlessness in Lung Cancer
Brief Title: Self-Management Intervention for Breathlessness in Lung Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Breathlessness Pilot
Record Dates: First submitted 2012-04-20; First posted 2012-04-26 (Estimated); Last update posted 2019-05-06 (Actual); Status verified 2019-05

CONDITIONS: Lung Cancer; Breathlessness
Keywords: Lung cancer; Breathlessness; Self-management
MeSH Terms: conditions — Lung Neoplasms; Dyspnea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Self-management Intervention (Experimental): Individual, face-to-face 7-session self-management intervention delivered by a specialist oncology nurse/clinical case manager as a home-based approach using a manual for each session.
  Interventions: Behavioral: Self-management Intervention
- Standard of care (Active Comparator): Patients in this condition will receive usual care as decided by their oncology clinic team or physician.
  Interventions: Behavioral: Self-management Intervention

INTERVENTIONS:
Behavioral: Self-management Intervention — Individual, face-to-face 7-session self-management intervention delivered by a specialist oncology nurse/clinical case manager as a home-based approach using a manual for each session. The intervention is delivered through scheduled home visits (7 sessions about one-hour in length), telephone coaching (2 sessions/week to reinforce use of strategies and for symptom monitoring: 15 minutes), and nurse moderated online peer chat or chat that is self-initiated at other times (7 weekly sessions about one hour in length).

SUMMARY:
The purpose of this study is to investigate the suitability and practicality of a coaching and support intervention in helping patients to use daily strategies for managing breathlessness. Also, the investigators will try to understand how useful it is in helping patients to reduce intensity of breathlessness and its impact their quality of life.

DETAILED DESCRIPTION:
Lung cancer is common worldwide and is a leading cause of death. Breathlessness (dyspnea or shortness of breath) is a highly prevalent clinical problem in lung cancer, developing early in 25-50% of patients due to advanced stage at presentation. It persists in 60% of survivors' post-lung resection and worsens with progressive disease with rates as high as 90% reported in the final months of life. Breathlessness is associated with a high degree of unpleasantness, negatively impacts on daily functioning, and multiple domains of quality of life, triggers fear and anxiety in patients and their family, and contributes to symptom specific and psychological distress. It is also costly to the health system as it contributes to urgent care use and hospitalization. The purpose of this pilot trial is to evaluate feasibility and acceptability of a self-management intervention for breathlessness in lung cancer.

ELIGIBILITY:
Inclusion criteria:

Eligible participants are women and men with lung cancer (stage I to IV) receiving chemotherapy and/or radiotherapy

1. Report breathlessness occurrence (any score >=3) on a Numerical Rating Scale (0-no breathlessness; 10 - worst breathlessness) during standardized routine distress screening and/or report breathlessness as a symptom to their health care provider
2. Normal cognitive function as measured by a score of <20 on the Short Orientation Memory Cognitive Test (SOMC)
3. ECOG performance score of 0 to 2
4. Estimated life expectancy of >3 months as per physician
5. Reside within a 45 kilometre driving radius of Princess Margaret Hospital
6. Oxygen saturation >90% at rest on room air or with oxygen
7. Available for 8 consecutive weeks of the study.

Exclusion criteria:

1. Patients who have received surgery alone as the primary treatment for lung cancer
2. Unstable acute asthma or left heart failure or coronary artery or valvular heart disease or neuromuscular disease
3. Inability to comply with the study protocol including completion of the questionnaires in English
4. Major psychiatric disorder identified by the physician.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2011-11-30 (Actual); Primary Completion 2015-12-30 (Actual); Study Completion 2015-12-30 (Actual)

PRIMARY OUTCOMES:
Perceived severity of breathlessness | 8 weeks
  Measured by Numeric Rating Scale for breathlessness intensity.
Affective distress of breathlessness | 8 weeks
  Measured by Distress of Breathlessness Numerical Rating Scale.
Dyspnea with activities of daily living and exercise | 8 weeks
  Measured by (a) Chronic Respiratory Questionnaire, (b) Medical Research Council Dyspnea Scale, and (c) BORG scale prior to, during, and at the end of the 6-Minute-Walk Test.

SECONDARY OUTCOMES:
Self-efficacy and mastery for managing breathlessness | 8 weeks
  Measured by (a) individual self-report items for "self-efficacy for managing shortness of breath" and "self-efficacy for exercise" from the toolkit of Stanford measures; (b) Chronic Respiratory Questionnaire - Mastery subscale; (c) adapted COPD Self-Efficacy Scale developed for this study.
Beliefs about breathlessness | 8 weeks
  Measured by Symptom Representation Questionnaire.
Adherence and Use of Self-Management Strategies | 8 weeks
  Measured using (1) Daily activity log of physical activity;(2)Seven-Day Physical Activity Recall tool (7-day PAR);(3) Cognitive Symptom Management Scale;(4) Daily tracking log of self-management strategies
Exercise capacity | 8 weeks
  Measured by 6-Minute Walk Test.
Psychological distress | 8 weeks
  Measured by the Hospital Anxiety and Depression Scale.
Quality of life | 8 weeks
  Measured by (a) Functional Assessment of Cancer Therapy - Lung (FACT-L); and, (b)Chronic Respiratory Questionnaire.
Health care utilization | 8 weeks
  Measured by three questions derived from the Stanford Self-Management Program Toolkit of Measures, regarding number of hospital days, emergency room visits, and visits to physicians related to their breathlessness.

CONTACTS AND LOCATIONS:
Overall Officials: Doris Howell, RN PhD, Principal Investigator — Princess Margaret Hospital, University Health Network
Locations (1):
- Princess Margaret Hospital/University Health Network, Toronto, Ontario, Canada